CLINICAL TRIAL: NCT02786316
Title: High Intensity Training in Patients With Non-Specific Chronic Low Back Pain: A Clinical Pilot Trial
Brief Title: High Intensity Training With Non-specific Chronic Low Back Pain
Acronym: LBP-HIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Annick Timmermans, prof. dr., Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBP-HIT-001
Record Dates: First submitted 2016-05-19; First posted 2016-06-01 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Experimental): Hit program for the rehabilitation of persons with nonspecific chronic low backpain
  Interventions: Other: HIT program
- Control group (Active Comparator): a conventional rehabilitation program for persons with nonspecific chronic low backpain
  Interventions: Other: conventional rehabilitation program

INTERVENTIONS:
Other: HIT program — HIT program for the rehabilitation of persons with NSCLBP
  Arms: intervention group
Other: conventional rehabilitation program — a conventional rehabilitation program in persons with NSCLBP
  Arms: Control group

SUMMARY:
Low back pain is a common disorder, occurring worldwide in both males and females in all age groups1. The prevalence is higher in females and the incidence peaks between 30 and 65 years. It is currently the most frequent musculoskeletal cause of functional disability and it has a major socio-economic impact on today's society. Although a small percentage of persons with low back pain can be diagnosed with a specific underlying cause, almost 90% of persons with low back pain present with symptoms of nonspecific origin. A part of these symptoms are only of short duration, but 23% of all people will develop nonspecific chronic low back pain (NSCLBP).

Exercise therapy (ET) is currently an important component in the treatment of NSCLBP. Previous studies analysed the effects of various modes of exercise therapy, such as motor control therapy, core stability training and aerobic conditioning training. However, therapy outcomes can be low, and guidelines in favour of using a specific program are contradictory. It thus still remains unclear which therapy modality is best suited. Furthermore, no recommendations are available about optimal training intensities during rehabilitation of persons with NSCLBP.

Since as well aerobic as muscular deconditioning are apparent in persons with chronic low back pain and improvements in overall physical fitness can affect therapy outcomes in this population, ET specifically focussing on physical fitness can be advocated for NSCLBP rehabilitation. High Intensity Training (HIT), has been promoted as an effective and efficient training method for improving physical fitness and health related parameters in healthy persons. Also, HIT resulted in successful reconditioning and improvement of functional and disease related outcomes in persons with other chronic diseases such as multiple sclerosis, heart failure, COPD and cardiometabolic diseases. Although some studies showed promising results for the effect of HIT on low back pain such as high intensity isolated, evidence is still scarce and study results are unclear because of methodological shortcomings.To evaluate HIT for the rehabilitation of persons with NSCLBP, a therapy program was developed consisting of high intensity interval cardio and high load whole body strength training.

The aim of this pilot study is 1) to evaluate the feasibility of a HIT program for the rehabilitation of persons with NSCLBP, and 2) to evaluate the effects of a HIT program on disease related outcomes and physical fitness compared to a conventional rehabilitation program in persons with NSCLBP.

ELIGIBILITY:
Inclusion Criteria:

1. medically diagnosed with non-specific chronic low back pain4,
2. over 18 years old,
3. able to understand Dutch (spoken and written).

Exclusion Criteria:

1. invasive surgery at the lumbar spine in the last 18 months (arthrodesis was excluded, microsurgery was allowed),
2. radiculopathy (uni- or bilateral),
3. co-morbidities: paresis and/or sensory disturbances by neurological causes, diabetes mellitus, rheumatoid arthritis, an increase of pain of 3 points with a result of > 8/10 on the Numeric Pain Rating Scale (NPRS) in the last 48 hours, pregnancy,
4. ongoing compensation claims and/or (work)disability > 6 months,
5. rehabilitation/exercise therapy program for LBP in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pain | day 1
  Numeric Pain Rating Scale (NPRS) The NPRS is a nominal scale on which the participant indicates the amount of pain he/she perceives at that current moment. It consists of a line indicating eleven successive scores (0-10), whereby score 0 means 'no pain' and score 10 means 'worst pain imaginable'. An improvement of 2 levels or more is accepted as clinically relevant
Pain | week 6
  Numeric Pain Rating Scale (NPRS) The NPRS is a nominal scale on which the participant indicates the amount of pain he/she perceives at that current moment. It consists of a line indicating eleven successive scores (0-10), whereby score 0 means 'no pain' and score 10 means 'worst pain imaginable'. An improvement of 2 levels or more is accepted as clinically relevant
Kinesiophobia | day 1
  Tampa Scale for Kinesiophobia (TSK) The TSK is an ordinal 17 item questionnaire that inventories pain-related fear of movement for persons with subacute and chronic low back pain or fibromyalgia41,42. A higher score relates to more pain-related fear.
Kinesiophobia | week 6
  Tampa Scale for Kinesiophobia (TSK) The TSK is an ordinal 17 item questionnaire that inventories pain-related fear of movement for persons with subacute and chronic low back pain or fibromyalgia41,42. A higher score relates to more pain-related fear.
physical disability | day 1
  Roland Morris Disability Questionnaire (RMDQ) The RMDQ is an ordinal 24 item questionnaire for evaluating the disability level of the patient with low back pain with regards to activities of daily living33,35. A higher score correlates to a higher level of disability and a change of 5 is the minimal clinically important difference36
physical disability | week 6
  Roland Morris Disability Questionnaire (RMDQ) The RMDQ is an ordinal 24 item questionnaire for evaluating the disability level of the patient with low back pain with regards to activities of daily living33,35. A higher score correlates to a higher level of disability and a change of 5 is the minimal clinically important difference36
Endurance capacity | day 1
  Endurance capacity test Endurance capacity is tested to volitional fatigue on an electronically braked bike ergometer (eBike Basic, General Electric GmbH, Bitz, Germany).
Endurance capacity | week 6
  Endurance capacity test Endurance capacity is tested to volitional fatigue on an electronically braked bike ergometer (eBike Basic, General Electric GmbH, Bitz, Germany).
Body composition | day 1
  Measured by Dual Energy X-ray absorptiometry (DEXA)
Body composition | week 6
  Measured by Dual Energy X-ray absorptiometry (DEXA)
weight | day 1
Weight | week 6
BMI (Body Mass Index) | day 1
BMI (Body Mass Index) | week 6

SECONDARY OUTCOMES:
physical activity | day 1
  Actigraph GT3X activity monitors Activity of the daily routine will be evaluated by means of wearing an accelerometer throughout 3 consecutive days. A schedule will be inventoried by the participant.
physical activity | week 6
  Actigraph GT3X activity monitors Activity of the daily routine will be evaluated by means of wearing an accelerometer throughout 3 consecutive days. A schedule will be inventoried by the participant.
disability in participation and quality of life | day 1
  Short Form Health Survey (SF-36)
disability in participation and quality of life | week 6
  Short Form Health Survey (SF-36)
Questionaire motivation and Therapy Adherence | day 1
Questionaire motivation and Therapy Adherence | week 6
  questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Verbrugghe, prof. dr., Study Chair — Hasselt University
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No